CLINICAL TRIAL: NCT05192928
Title: Understanding the Feasibility of Ripple Health Smart Pill Caps in Clinical Settings, and the Devices' Effects on Medical Interventions.
Brief Title: Feasibility of Ripple Health Smart Pill Caps in Clinical Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manan Shukla (Industry)
Responsible Party: Sponsor-Investigator, Manan Shukla, Founder, Ripple Health
Organization: Ripple Health (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1280044
Record Dates: First submitted 2021-12-17; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Chronic Disease; Asthma
Keywords: Compliance; Interventions; Feasibility
MeSH Terms: conditions — Chronic Disease; Asthma; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- All Patients using the Ripple Health Smart Pill Cap (Experimental): In this single-arm trial, all patients will be using the Ripple Health Smart Pill Cap as a method of medication administration
  Interventions: Device: Ripple Health Smart Pill Cap

INTERVENTIONS:
Device: Ripple Health Smart Pill Cap — The device is a smart medical device created to allow physicians to have better access to patient compliance data, and intervene on the patient's health through the use of a text message, phone call, or email.
  Other Names: Ripple Health Smart Pill Bottle

SUMMARY:
The purpose of this research is to determine whether Ripple Health Smart Medicine Bottle Caps can allow for better interface medication administration than traditional pill bottles. A secondary goal of the study is to determine whether the smart medication caps can allow the physician to intervene in the patient's health regimen when necessary. This occurs when the patient does not take medication for reasons such as the painful side effects of the medication, or the high cost of the medication itself. By intervening, a physician can therefore help increase patient adherence, and improve transparency between the patient and the physician

The bottle cap is in essence a pill bottle that contains circuitry in the cap of the bottle, which sends data to a physician over a wifi network. Once the patient opens the pill bottle, sensors inside the bottle cap will trigger, and send data to the web server indicating that the patient has taken the medication(we are assuming that the patient takes the medication if he/she opens the pill bottle). The server will then add this data into a database that is available to the physician to view. In this study, the proposed use of this pill bottle is as a simple medication container that gets opened when the patient needs to take his/her medication.

DETAILED DESCRIPTION:
Approximately 133 million or six out of ten patients are affected by at least one chronic disease such as heart disease, stroke or diabetes (National Health Council). Although these diseases can be treated easily using medications, millions of adults die inside the hospital room due to chronic complications. This is due to a problem known as Medical Non-adherence, in which millions of patients do not take their medication as prescribed by the physician. This inhibits the physician's ability to properly treat their patients, leading to a poor patient outcome. Such an issue has affected almost every aspect of healthcare, from avoidable hospitalization to insurance wastes. At the same time, clinical trial results also tend to be skewed because the variable of adherence is not controlled.

The Ripple Health patented smart pill dispenser was therefore created as one of the first objective healthcare technologies that can send real-time patient adherence information to the physician and pharmacist through an IoT Cloud system. Not only can the device provide useful insights to pharmacies, physicians and the patient's loved ones, but it can also save billions of dollars lost by insurance companies, hospitals and the Center of Medicare Services by reducing avoidable hospitalizations and allowing the patient to remain on their treatment regimen. Finally, by implementing such a technology in clinical experiments, the probability of skewed results will decrease as medical adherence in a clinical field will be more controlled.

At the same time, the Ripple Health dispenser is also affordable, with a cost of approximately three dollars mass-produced. By becoming extremely cost effective, not only will most patients be able to afford it, but this device will be widely available to patients around the country at a negligible price.

The purpose of this research is to determine whether Ripple Health Smart Medicine Bottle Caps can allow for better interface medication administration than traditional pill bottles. A secondary goal of the study is to determine whether the smart medication caps can allow the physician to intervene in the patient's health regimen when necessary. This occurs when the patient does not take medication for reasons such as the painful side effects of the medication, or the high cost of the medication itself. By intervening, a physician can therefore help increase patient adherence, and improve transparency between the patient and the physician

The bottle cap is in essence a pill bottle that contains circuitry in the cap of the bottle, which sends data to a physician over a wifi network. Once the patient opens the pill bottle, sensors inside the bottle cap will trigger, and send data to the web server indicating that the patient has taken the medication(we are assuming that the patient takes the medication if he/she opens the pill bottle). The server will then add this data into a database that is available to the physician to view. In this study, the proposed use of this pill bottle is as a simple medication container that gets opened when the patient needs to take his/her medication.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the clinic above the age of 18 with the ability to consent and have a prescribed medication from the clinic will be asked to participate in the study. All patients also must be proficient in English.
* Patients who are minors are required do have at least 1 capable guardian/parent who will be administering the medication and using the pill bottle.

This will be determined by the physician, as he has seen such a patient in the past. The physician will determine whether the patient has a physical or mental condition and thus will be excluded from the study.

* The parent of the minor must also be mentally and physically capable of opening the pill bottle.
* Patients are also required to have wifi-connectivity in order to consent.

Exclusion Criteria:

* All subjects in the study must be above the age of 18- whether they are the patients themselves, or the parents of the patients. All age related criteria about the patient can be determined from an EHR service that is already being used in the clinic
* Patients who cannot use the bottle due to a physical(cannot open the bottle) or mental condition will not be allowed to participate in the study. This will be determined by the physician, as he has seen such a patient in the past. The physician will determine whether the patient has a physical or mental condition and thus will be excluded from the study.
* Patients above 18 who are unable to consent will be excluded from the study. The ability to consent will be determined through the physician, who will decide whether the patient is able to consent to the study. The physician, who has worked with the patient significantly in the past, will be able to determine whether the patient is able to consent to the study.
* Minors whose guardian/parent is unable to consent will be excluded from the study. This will be determined by the physician, as he has seen such a patient in the past. The physician will determine whether the patient has a physical or mental condition and thus will be excluded from the study. The parents of the minors must also be able to physically open the pill bottle.
* Minors who are mentally and physically incapable will be excluded from the study. This will be determined by the physician, as he has seen such a patient in the past. The physician will determine whether the patient has a physical or mental condition and thus will be excluded from the study.
* Patients without wifi connectivity will be excluded from the study. We can determine patients who have wifi-connectivity by asking the patient if he/she has connectivity in his/her residence. Patients who have limited English proficiency will be excluded from the study. This can be determined through conversation with the patient. If the patient shows signs of a limited English proficiency, the patient will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Amount of provider interventions done per patient | 1 month
  Measures the total amount of provider interventions when the patient was non-compliant.
Total number of malfunctions present throughout the trial | 1 month
  Measures the total amount of malfunctions each device had throughout the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Manan Shukla, Principal Investigator
Locations (4):
- United States (4):
  - Allergy Asthma Sleep Center, Astoria, New York
  - Allergy Asthma Sleep Center, Brooklyn, New York
  - Allergy Asthma Sleep Center, New York, New York
  - Allergy Asthma Sleep Center, Staten Island, New York

IPD SHARING:
Plan to Share IPD: No